CLINICAL TRIAL: NCT02633436
Title: Research on the Role of the Amino Acid Transporter SLC1A5 in the Development of Esophageal Cancer
Brief Title: Research on the Role of SLC1A5 in the Development of Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fourth Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Liuzhou Maternity and Child Healthcare Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PJK201518
Record Dates: First submitted 2015-12-06; First posted 2015-12-17 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Esophageal Cancer; Amino Acid Transport Disorder
Keywords: esophageal cancer; SLC1A5
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — Tissue specimens of esophageal cancer patients will be collected and stored in liquid nitrogen after operations
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cancer tissues: SLC1A5 expression of esophageal cancer tissues from patients
  Interventions: Other: SLC1A5 expression
- paired adjacent tissues: SLC1A5 expression of paired adjacent esophageal tissues from patients
  Interventions: Other: SLC1A5 expression

INTERVENTIONS:
Other: SLC1A5 expression — To observe the expression of SLC1A5 by immunohistochemistry and WesternBlot analysis.

SUMMARY:
To explore the significance of Solute Carrier Family 1 Member 5 (SLC1A5) in the occurrence of esophageal cancer, by comparing the expression of SLC1A5 between esophageal cancer tissues and adjacent tissues.

DETAILED DESCRIPTION:
This will be an observational study. The investigators will aim to enroll 100 male and female adult patients (aged 18 years and over) of all ethnicities/races, who have been referred to the Fourth Affiliated Hospital of Guangxi Medical University for esophageal cancer.

The investigators will be using a standardized data collection form. This is an observational study in which standard of care will be practiced and the patients are not placed at additional risk from participating in this study. However, as the investigators are collecting data prospectively, all participants will sign consent. An attempt will be made to see if there is a correlation between the expression of SLC1A5 with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven esophageal cancer;
2. Age ≥18 years;
3. All patients must sign consent forms voluntarily;

Exclusion Criteria:

1. Inability to obtain histologic proof of malignancy.
2. Age <18 years;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven esophageal cancer
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
optical density (ODs) of each slice by immunohistochemistry assay | within one year (plus or minus 1 month) after surgery
  For immunohistochemistry assay： Briefly, the samples will be cut into slices, which will be stained with standard steps. Finally, three high power fields will be randomly selected from each slice and the average optical density (OD) will be measured in each field.

SECONDARY OUTCOMES:
SLC1A5 expression detected by WesternBlot | within one year (plus or minus 1 month) after surgery
  Western blot assay will be done by comparing the intensity of bands. To start with, xray film will be scanned on a flat-bed scanner. Then the grayscale image will be analyzed with software. Finally the Gray Value of each band will be obtained for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcheng Wei, Principal Investigator — Guangxi Medical University Institutional Review Board
Locations (2):
- China (2):
  - Liuzhou Maternity and Child Healthcare Hospital, Liuchow, Guangxi
  - The Fourth Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi

IPD SHARING:
Plan to Share IPD: Undecided